CLINICAL TRIAL: NCT02999763
Title: Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction
Brief Title: SlimShape Device for Abdominal Fat and Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF22621
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Fat Disorder
Keywords: lipolysis; fat reduction; circumference reduction
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abdominal fat reduction treatment (Experimental): SlimShape treatments will be administered for up to 3 sessions to the abdomen of all study participants.
  Interventions: Device: SlimShape

INTERVENTIONS:
Device: SlimShape — SlimShape radiofrequency treatment to the abdomen

SUMMARY:
Prospective, one-arm, baseline-controlled, clinical study for the evaluation of the SlimShape device for non-invasive abdominal fat and circumference reduction.

Study subjects will undergo SlimShape treatments on the abdominal area.

DETAILED DESCRIPTION:
The objective of this trial is to evaluate the safety and efficacy of the SlimShape device utilizing the SlimShape Applicator Belt for abdominal non-invasive fat and circumference reduction. Eligible subjects will receive up to 3 bi-weekly treatments (2 weeks interval) with the SlimShape device utilizing the SlimShape Applicator Belt according to the study protocol.

The subject will return for 3 follow up visits: four weeks (4wk FU), eight weeks (8wk FU) and 12 weeks (12wk FU) after the last treatment.

Each subject will be enrolled for total expected study duration of up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects, ≥18 and ≤60 years of age at the time of enrollment
3. Fitzpatrick Skin Type I to VI
4. BMI interval: 18.5 ≤ BMI ≤ 30 (normal to overweight, but not obese).
5. If female, not pregnant, lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
6. In addition, negative urine pregnancy test as tested before each treatment and at the last visit for women with childbearing potential (e.g. not menopause).
7. General good health confirmed by medical history and skin examination of the treated area.
8. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
9. Willing to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
10. Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations.

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
2. Current hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone
6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction
7. Previous body contouring procedures in the treatment area within 12 months
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
9. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity)
10. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
11. Allergy to any component of the lotion (VelaSpray Ease) used in this study
12. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
13. Very poor skin quality (i.e., severe laxity)
14. Abdominal wall diastasis or hernia on physical examination
15. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
16. Obesity (BMI > 30)
17. Childbirth within the last 12 months or breastfeeding women. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
18. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months)
19. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration).
20. Participation in another clinical study involving same anatomical areas within the last 6 months (or 30 days in case different anatomical areas were treated in previous trial/s).
21. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruthie Amir, MD, Study Director — Syneron Medical
Locations (4):
- United States (4):
  - Laser & Skin Surgery Medical Group, Inc, Sacramento, California
  - Syneron Candela Institute for Education Clinic, Wayland, Massachusetts
  - Union Square Laser Dermatology, New York, New York
  - Laser & Skin Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adatto MA, Adatto-Neilson RM, Morren G. Reduction in adipose tissue volume using a new high-power radiofrequency technology combined with infrared light and mechanical manipulation for body contouring. Lasers Med Sci. 2014 Sep;29(5):1627-31. doi: 10.1007/s10103-014-1564-x. Epub 2014 Apr 1. PMID 24687404

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated and Untreated Abdomen: Circumference and fat thickness reduction of abdomen after SlimShape treatments (three treatments with SlimShape RF based device)
Period: Overall Study
Arm/Group | Treated and Untreated Abdomen
Started | 70
Completed | 58
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- Treated and Untreated Abdomen: Circumference and fat thickness measurements of abdomen before after SlimShape treatments of the same subjects
Arm/Group | Treated and Untreated Abdomen
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 61
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 70
Fat Thickness [Mean (Standard Deviation); unit: millimeter] | 22.83 (7.22)
Circumference [Mean (Standard Deviation); unit: centimeter] | 91.64 (7.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat Thickness at Final Follow-up Compared to Baseline
Description: Abdominal fat change, measured by ultrasound, post SlimShape treatments at 12 weeks follow-up (12wk FU) compared to baseline
Time Frame: Baseline and 12 weeks follow-up
Population: 58 participants analyzed at 12 week FU (12 subjects lost to follow-up at final visit)
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Treated Abdomen: Subjects treated on the abdomen with SlimShape RF treatments
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 58
millimeters | -1.76 (1.4)

2. Secondary Outcome: Change in Fat Thickness After Treatments Compared to Baseline
Description: Abdominal fat change, measured by ultrasound, post SlimShape treatments at 4 and 8 weeks follow-up after final treatment compared to baseline
Time Frame: Baseline and 4 and 8 weeks follow-up
Population: 63 participants attended the 4 week FU (5 dropped and 2 missed the visit), 59 participants attended the 8 week FU (10 dropped and 1 missed the visit)
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 70
millimeters
  Fat thickness change at 4 week FU: number analyzed (Participants) | 63
  Fat thickness change at 4 week FU | -0.51 (2.2)
  Fat thickness change at 8 week FU: number analyzed (Participants) | 59
  Fat thickness change at 8 week FU | -1.33 (2.3)

3. Secondary Outcome: Change in Abdominal Circumference After Treatments Compared to Baseline
Description: Change in abdominal circumference, measured by calibrated measuring tape, at 4, 8 and 12 weeks follow-up (after final treatment) compared to baseline
Time Frame: At 4 weeks, 8 weeks and 12 weeks follow-up (post last treatment)
Population: 63 participants attended the 4 week FU (5 dropped and 2 missed the visit), 59 participants attended the 8 week FU (10 dropped and 1 missed the visit), 58 participants attended the 12 week FU (12 Subjects dropped)
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 70
centimeter
  Abdominal circumference change at 4 week FU: number analyzed (Participants) | 63
  Abdominal circumference change at 4 week FU | -0.53 (2.6)
  Abdominal circumference change at 8 week FU: number analyzed (Participants) | 59
  Abdominal circumference change at 8 week FU | -0.53 (2.6)
  Abdominal circumference change at 12 week FU: number analyzed (Participants) | 58
  Abdominal circumference change at 12 week FU | -0.78 (2.7)

4. Other Pre Specified Outcome: Number of Treatments Where Participants Reported Having "Mild", "Moderate" or "Severe" Response
Description: Discomfort and immediate response will be assessed immediately after each treatment using the Post Treatment Immediate Response severity scale (Absent/none, Mild, Moderate and Severe). The values in the data table reflect the number of participants who had discomfort during treatment or immediate response after treatment (reported as having "Mild", "Moderate" or "Severe" )
Time Frame: First, second and third treatments, Weeks 0 to 4
Population: 70 participants attended the first treatment, 67 participants attended the second treatment (2 dropped and 1 missed treatment) and 65 participants attended the third treatment (3 dropped and 2 missed treatment), therefore overall 202 treatments conducted during the study.
Measure: Count of Units; unit: Overall Treatments
Units Other Than Participants: Overall Treatments
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 70
Number analyzed (Overall Treatments) | 202
Overall Treatments
  The rate of erythema after treatment | 199
  The rate of edema after treatment | 84
  The rate of hematoma / purpura after treatment | 11
  The rate of petechiae after treatment | 35
  The rate of pain after treatment | 19

ADVERSE EVENTS:
Time Frame: Subjects were assessed and followed up for adverse events at each treatment (3 treatment at 2 weeks interval) and at 4 weeks, 8 weeks and 12 weeks after the SlimShape treatment
Arm/Group | Treated Abdomen
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 10/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Abdomen (N=70)
Blisters (Skin and subcutaneous tissue disorders) | 7 (7) — All blisters recovered during study period
Vesicles (Skin and subcutaneous tissue disorders) | 1 (2) — Vesicles on the left and right side of the abdomen
Discoloration (Skin and subcutaneous tissue disorders) | 1 (1) — Mild discoloration
firm mass (Skin and subcutaneous tissue disorders) | 1 (1) — small 1x1 cm firm mass

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT02999763/Prot_SAP_000.pdf